CLINICAL TRIAL: NCT01279499
Title: Propofol Versus Sevoflurane as Sole Anesthetic Agent in Gastric By-Pass Surgery for Morbid Obesity: A Prospective Randomized Clinical Trial
Brief Title: Sevoflurane Versus Intravenous Anaesthetic Agents in Morbid Obese Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Patras (Other)
Responsible Party: Kriton Filos, University of Patras, Departement of Anesthesiology and Critical Care Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: sevoflurane-propofol-obesity
Record Dates: First submitted 2011-01-11; First posted 2011-01-19 (Estimated); Last update posted 2011-01-20 (Estimated); Status verified 2010-03

CONDITIONS: Morbid Obesity
Keywords: Morbid obesity; Sevoflurane; Propofol; Remifentanyl; BIS; Cardiovascular stability; Recovery scores; Drug consumption
MeSH Terms: conditions — Obesity, Morbid | interventions — Sevoflurane; Propofol; Remifentanil; halofantrine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- SEVO group (Active Comparator): Anaesthesia will be induced with IV Propofol (2 mg/kg TW [TW = ideal body weight, IBW + 0.4 * difference to the excess weight]), Remifentanyl (1 μg/kg IBW) and succinylcholine (1mg/kg IBW).Intraoperatively Sevoflurane will be guided by a target end tidal concentration 1 - 2 MAC .Every rise of BP or HR > 15% of baseline will be followed by a bolus SEVO inhalation 8% MAC for 2 minutes.If the positive sympathetic response persists, then Nifedipine 10 mg will be administered sublingual, if HR < 70/ minute, and Diltiazem 10-20 mg IV will be administered if HR > 70/ minute, followed by esmolol administration if response to diltiazem is unsatisfactory. The duration and frequency of positive sympathetic stress responses that required pharmacologic intervention will be recorded.
  Interventions: Drug: Sevoflurane
- SEVO-BIS group (Active Comparator): Anaesthesia will be induced with IV Propofol (2 mg/kg TW [TW = ideal body weight, IBW + 0.4 * difference to the excess weight]), Remifentanyl (1 μg/kg IBW) and succinylcholine (1mg/kg IBW).Intraoperatively Sevoflurane will be guided by a target BIS of 40 - 50 .Every rise of BP or HR > 15% of baseline will be followed by a bolus SEVO inhalation 8% MAC for 2 minutes. If the positive sympathetic response persists, then Nifedipine 10 mg will be administered sublingual, if HR < 70/ minute, and Diltiazem 10-20 mg IV will be administered if HR > 70/ minute, followed by esmolol administration if response to diltiazem is unsatisfactory. The duration and frequency of positive sympathetic stress responses that required pharmacologic intervention will be recorded.
  Interventions: Drug: Sevoflurane
- Propo- Remi group (Active Comparator): General Anaesthesia (GA) will be induced with a continuous IV Propofol (P) infusion (21mg/kg TBW for 5 min, 12 mg/kg TBW for 10 min and then 6 mg/kg TBW), followed by an IV bolus of Remifentanyl (R, 1 μg/kg IBW) and succinylcholine (1mg/kg IBW). GA will be maintained with continuous intravenous administration of P at 150-300mcg/kg/min (doses based on ideal body weight).
  Every rise of BP or HR > 15% of baseline will be followed by a R bolus IV (1 μg/kg IBW) and increase in the continuous infusion rate of R to 1.0 μg/kg/min . If HR < 70/ minute, and Diltiazem 10-20 mg IV will be administered if HR > 70/ minute, followed by esmolol administration if response to diltiazem is unsatisfactory. The duration and frequency of stress responses that required intervention is recorded.
  Interventions: Drug: Propofol- Remifentanyl
- Propo-Remi-BIS group (Active Comparator): General Anaesthesia (GA) will be induced with a continuous IV Propofol (P) infusion (21mg/kg TBW for 5 min, 12 mg/kg TBW for 10 min and then 6 mg/kg TBW), followed by an IV bolus of Remifentanyl (R, 1 μg/kg IBW) and succinylcholine (1mg/kg IBW). GA will be maintained with continuous intravenous administration of P at 150-300mcg/kg/min (IBW).
  The depth of anesthesia will be adjusted to accomplish a BIS score 40 -50. If BP or HR is > 15% of baseline will a bolus of R IV (1 μg/kg IBW) will be given and an the infusion rate of R will be increased to 1.0 μg/kg/min . If this response persists and HR < 70/ min, Nifedipine 10 mg will be given s.l. and if HR > 70/ min Diltiazem 10-20 mg IV will be given, followed by esmolol infusion if no response is observed.
  Interventions: Drug: Propofol, Remifentanyl

INTERVENTIONS:
Drug: Sevoflurane — Intraoperatively Sevoflurane will be guided by a target end tidal concentration 1 - 2 MAC .Every rise of BP or HR > 15% of baseline will be followed by a bolus SEVO inhalation 8% MAC for 2 minutes
  Other Names: Sevoflurane , Abbott
  Arms: SEVO group
Drug: Sevoflurane — Intraoperatively sevoflurane will be guided by a target BIS of 40 - 50. If a positive sympathetic response occured (an elevation of the HR and/or MAP greater than 15% above baseline) a bolus SEVO 8 MAC will be administered for 2 minutes.
  Other Names: Sevoflurane, Abbott and BIS, Aspect Medical Systems, USA
  Arms: SEVO-BIS group
Drug: Propofol- Remifentanyl — Anaesthesia will be induced with a continuous IV Propofol infusion (21mg/kg TBW for 5 min, 12 mg/kg TBW for 10 min and then 6 mg/kg TBW), followed by an IV bolus of Remifentanyl (1 μg/kg IBW) and succinylcholine (1mg/kg IBW).General anesthesia will be maintained with continuous intravenous administration of Propofol at 150-300mcg/kg/min (doses based on ideal body weight).
  Every rise of BP or HR > 15% of baseline will be followed by a Remifentanyl bolus IV (1 μg/kg IBW) and increase in the continuous infusion rate of Remifentanyl from 0.1 to 1.0 μg/kg/min
  Other Names: Propofol, Diprivan, Fresenius; Remifentanyl, Ultiva, GlaxoSmithKline
  Arms: Propo- Remi group
Drug: Propofol, Remifentanyl — Anaesthesia will be induced with a continuous IV Propofol infusion (21mg/kg TBW for 5 min, 12 mg/kg TBW for 10 min and then 6 mg/kg TBW), followed by an IV bolus of Remifentanyl (1 μg/kg IBW) and succinylcholine (1mg/kg IBW). General anesthesia will be maintained with continuous intravenous administration of Propofol at 150-300mcg/kg/min (ideal body weight).
  The depth of anesthesia will be adjusted so as to accomplish a BIS score between 40 and 50 Every rise of BP or HR > 15% of baseline will be followed by a Remi bolus IV (1 μg/kg IBW) and increase in the continuous infusion rate of Remi from 0.1 to 1.0 μg/kg/min
  Other Names: Propofol, Fresenius, BIS, Aspect Medical Systems, USA
  Arms: Propo-Remi-BIS group

SUMMARY:
The objective of this prospective randomized clinical study was to compare anesthesia, in morbidly obese patents (BMI >50) who underwent BPD-RYGBP with either sevoflurane or propofol with remifentanyl.

DETAILED DESCRIPTION:
This is a prospective double blind randomized controlled trial. The patients will be assigned to one of 4 groups (gr): (1) SEVO group, guided by a target end tidal concentration 1 - 2 MAC and modified according to the haemodynamics (BP, HR) of the patients using a bolus inhalation (4 MAC), (2) SEVO-BIS group, using SEVO to a target BIS of 40 - 50, (3) PROPO-REMI and (4) PROPO-REMI-BIS groups accordingly. In groups 1 and 2, anaesthesia will be induced with IV PROPO (2 mg/kg TW [TW = ideal body weight, IBW + 0.4 * difference to the excess weight]), REMI (1 μg/kg IBW) and succinylcholine (1mg/kg IBW). In groups 3, 4 anaesthesia will be induced with a continuous IV PROPO infusion (21mg/kg TW/h for 5 min, 12 mg/kg TW/h for 10 min and then 6 mg/kg TW/h), followed by an IV bolus of REMI and succinylcholine as above. Every rise of BP or HR > 15% of baseline will be followed by a bolus SEVO inhalation in grs 1 and 2 or REMI bolus IV (1 μg/kg IBW) and increase in the continuous infusion rate of REMI from 0.1 to 1.0 μg/kg/min in groups 3 and 4. An epidural catheter will be placed prior to induction for postoperative analgesia only. Intraoperative BP and HR, anaesthetic consumption, recovery scores (Aldrete, Chung, White) and anaesthesia cost will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 yrs
* BMI>50 kg/m2
* Written consent for the participation in the study

Exclusion Criteria:

* History of significant cardiac disease, (aortic stenosis, angina, CHF or previous cardiac or intrathoracic operations)
* Significant renal dysfunction (serum creatinine>1.8 mg/dl)
* Significant liver dysfunction (evidenced by abnormal LFTs)
* History of hyper or hypothyroidism
* History of psychiatric or neurologic disorders
* Recall during general anesthesia
* Substance abuse (alcohol or other drugs)
* Counter-indications of placement of thoracic epidural catheter( previous spine surgery or coagulation abnormalities )
* Refusal to participate in the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-06 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of perioperative haemodynamic measurements (HR, MAP), recovery scores (Aldrete, White,Chung) | 5 min after induction, 1 hour after induction, end of the surgery, 2 hours postoperatively

SECONDARY OUTCOMES:
Drug Consumption, Drug Cost. | End of the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Athina Siampalioth, MD, Principal Investigator — University of Patras, Departement of Anesthesiology and Critical Care Medicine; Kriton Filos, Professor, MD, PhD, Study Chair — University of Patras, Departement of Anesthesiology and Critical Care Medicine
Locations (1):
- University Hospital of Patras, Departement of Anesthesiology and Critical Care Medicine, Pátrai, Achaia, Greece